CLINICAL TRIAL: NCT05684432
Title: Frequency and Classification of Radiation-induced Diarrhoea in Patients with Prostate and Rectal Cancer During Curative External Radiotherapy
Brief Title: Radiation-induced Diarrhoea During Curative EBRT of Prostate and Rectal Cancer
Acronym: PRECANU
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Mette Overgaard Holm, PhD student, Aalborg University Hospital
Other Study IDs: N-20210040
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-02

CONDITIONS: Radiation-induced Diarrhoea in Prostate and Rectal Cancer
Keywords: Acute radiation-induced diarrhoea; Curative EBRT; Prostate cancer; Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Faecal samples and blood during RID in a sub cohort of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prostate and rectal cancer patients: Curative EBRT
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Approx. 80% of patients with prostate and rectal cancer who receive radiation therapy (RT) experience acute radiation-induced diarrhea (RID). RID has major impact on patients' quality of life, can lead to pause or early termination of RT and chronic diarrhea. RID is poorly described with few details of type and severity of RID in clinical practice and in the literature. We are conducting an observational study in patients in patients who receive curative EBRT radiation for prostate and rectal cancer to uncover the frequency and classifications of RID.

DETAILED DESCRIPTION:
1. Background Prostate and rectal cancer are among the most common cancer types in Denmark and make up the majority of patients who receive curative radiation therapy of the small pelvis. A well-known side effect of external beam radiation therapy (EBRT) to the pelvis is radiation-induced diarrhoea (RID). When ionising radiation is given to the patient, both tumour and the surrounding cells are damaged. Thus, irradiating prostate and rectal cancer will inevitably lead to the damage of the nearby gut mucosa cellular components. This cellular damage is causing the RID. RID is reported as the problem with the greatest impact on health-related quality of life (QoL) and social behaviour.

   Up to approx. 70% of patients who receive pelvic radiation experience acute RID. It usually occurs two weeks after start of EBRT and peaks during 4-5 weeks. Acute RID may cease a few weeks after the end of EBRT but increases the risk of developing chronic RID.

   Recently, a systematic Cochrane review reveals low evidence for dietary interventions in RID due to few studies and low scientific quality. A serious drawback of the Cochrane review was that it included studies prior of 2005, with radiotherapy given both pre- and post-surgery, as well as with radiotherapy techniques resulting in higher doses to the normal tissue. It is well known that the volume of the radiation field greatly impacts the severity of RID and newer radiation techniques allow smaller volume fields.

   There is a lack of consensus about how acute RID is reported, such as definition of RID (frequency), classification and the changes during EBRT. There is also a lack of knowledge of changes in microbiomes which can contribute to RID. The role of dietary intervention during EBRT could also influence RID.
2. Aim The aim of this prospective observation study is to investigate the frequency, severity and changes of acute RID in patients with prostate and rectal cancer as well as the role of nutrition and changes in microbiome during curative EBRT.
3. Method This is an observational multicenter study of acute RID in patients with prostate and rectal cancer during curative EBRT. The study will take place in parallel with the patients' EBRT, which is ongoing on weekdays over 39 days for patients with prostate cancer and 28 days for patients with rectal cancer.

Study procedure Candidates will be identified according to the inclusion and exclusion criteria. The patients will be informed orally and in written form by a doctor or project nurse at the first oncology appointment.

The observations will start at baseline and concomitant with EBRT. All examinations and observations will be carried out in parallel with the patient's EBRT.

Data collection

1. Patient data: Civil status, age, sex, comorbidities, smoking, histopathology data: Primary diagnosis, date, stage, Electronic patient's record (EPR) 2. Treatment data: Treatment start and end date, fractionation and total dose (Gy), field size and anatomical location, EPR 3. Clinical examinations: ECOG performance status, body weight, height, rectal exploration, rectal haemorrhage or mucus, bloating, flatulence, obstipation, abdominal pain or tenesmus, faecal or urine incontinence, EPR, Common Terminology Criteria for Adverse Events (CTCAE) 4. Medication: Anti-diarrhoeal medication, laxatives, antibiotics, opioids, EPR 5. Frequency and classification of RID, body weight, Bristol Stool Scale and patient reported stool diary 6. Nutrition screening: Nutrition-related symptoms, dietary intake development, PG-SGA-short form 7. Dietary assessment: 3-day food records, online food database (Vitakost, 2006-2018, Denmark 8. Patient's physical activity, International Physical Activity Questionnaire (IPAQ-short form) 9. Quality of life (QoL), EORTC QLQ-C30, EORTC QLQ-PRT20 questionnaires 10. Biochemistry: Routinely blood samples collected at baseline will be obtained, EPR (biochemical record) 11. Faecel samples only for patients treated in Aalborg: F-calprotectin, short chain fatty acids. Samples will be frozen for subsequent microbial analysis, EPR (microbiological record)

4. Statistical considerations It is expected to include at least 100 patients during the inclusion period from 1 June 2022 to 31 December 2023. We expect to find above 30% of the patients with acute RID, why the required number of patients is estimated as above. The data are processed descriptive, as current numbers and percentages.

Uni- and multivariate analyses will be conducted using the Stata software, version 16 (StataCorp, LLC, TX, USA).

5. Subjects Patients with prostate and rectal cancer patients commenced to start curative EBRT, referred to the oncology department at Danish hospitals participating in the study will be consecutively screened for study eligibility according to the inclusion and exclusion criteria.

1. Inclusion criteria

   1. Histopathologically verified prostate or rectal adenocarcinoma 2. Commenced to start curative EBRT to the pelvis, with or without chemotherapy or with or without androgen deprivation therapy (ADT) 3. Performance status 0-1 4. ≥ 18 years of age 5. Understanding and acceptance of written and orally informed consent in Danish
2. Exclusion criteria

   1. Earlier treated with EBRT or other type of radiation to the pelvis
   2. History of diagnosed inflammatory bowel disease
   3. Colostomy
   4. Pregnancy

   6. Risks, side effects and disadvantages in short and long term This observational study does not include any risks for the included patients. Their treatment will be carried out as standard of care. Disadvantages are only related to answering the questionnaires and extra blood-samples and for Aalborg-patients also the collection of stool-samples.

   7. Information from patient records

   The following data will be registered:

   Civil status, age, sex, smoking, comorbidities, histopathologal data: primary diagnosis, date, stage.

   Treatment start and end date, fractionation and total dose (Gy), field size and anatomical location.

   Clinical examinations: ECOG performance status, rectal exploration, rectal haemorrhage or mucus, bloating, flatulence, obstipation, abdominal pain or tenesmus, faecal or urine incontinence.

   8. Data collection The tools (PG-SGAshort form, IPAQ short form, EORTC QLQ-C30 and EORTC QLQ-PRT20) will be sent to the patient's email address or security electronic mailbox (e-Boks) via RedCAP. Patient's responses will be registered directly in RedCAP.

   Patient reported stool diary and 3-day food records will be handed out in paper versions at the 1st visit at the radiation center. These paper versions will be returned to the primary investigator via franked envelopes and the data recorded will be registered in RedCAP. Data collected will be handled according to the Danish law of data protection and Personal Data Act. It is the responsibility of the principal investigator to ensure that the rules and regulations of data collection and storage comply with the Personal Data Act.

   9. Data storage The patient's personal identification/CPR number will be removed and replaced by a code number.

   All data will be stored in the MM-ICI-ABX research database in the system of the Research Electronic Data Capture (REDCap) at the clinical research unit, Dept. of Oncology, Aalborg University Hospital, the North Region of Denmark.

   10. Data protection All data stored in the REDCap research data MM-ICI-ABX will be handled according to the rules of Good Clinical Research Practice (27). The research database will be stored at the Clinical Research Unit, Dept. of Oncology, Aalborg University Hospital and owned by the Northern Region of Denmark. The password will be established for the principal investigator only (Mette Overgaard Holm). The members of the project group will handle the data according to the Danish laws of personal data protection. The patient's personal identification number will be removed and replaced of a code number (anonymisation). The key document with information on both personal ID and code number will be deposited at the clinical research unit project secretary according to GDPR and the Danish laws of personal data protection.

   11. Data deletion All data in this study will be deleted 5 years after publication of all results.

   12. Collaboration agreement Collaboration agreement will be made between the principal investigator in the North Denmark Region and the participating local investigators of the actual regions of Denmark (The Capital Region of Denmark, Region Zealand and South Denmark Region).

   The study will be performed between the North Denmark Region, the Capital Region of Denmark, region Zealand and South Denmark Region. The study will be designed by all responsible parts.

   13. Economy The initiative for this project was taken by the project group, employed at Aalborg University Hospital and Clinical Institute, Aalborg University. Participants in the project group are financed (partial or completely) through their employment at Aalborg University Hospital and Clinical Institute, Aalborg University.

   Funding of 320,000 DKK has been obtained from the Clinical Institute, Aalborg University (research fund, U. Falkmer) and from the Region North Denmark of 86,000 DKK (research fund, M.O. Holm), as well as 191,850 DKK from the Danish Comprehensive Cancer Center (DCCC) and will be used for salary for the PhD student (Mette Overgaard Holm), statistician, as well as a coordinative staff from each participating radiation therapy center. There is no economic benefit for neither the participating departments nor the hospital employees.

   The funders have no role in study design, data collection and analysis, and decisions to publish, or preparation of the manuscript.

   14. Compensation and/or other benefits to the subjects The patients will not be offered any financial compensation or other benefits due to study participation, nor travel expenses.

   Patients participating in the study are covered by national regulation.

   15. Publication The results regardless of positive, negative, and inconclusive character will be published in international peer reviewed scientific journals and in the PhD thesis of Mette Overgaard Holm.

   16. Science ethics section All patients included in the study have signed their information used for this clinical research project. The study is initiated as an academic protocol of the project group. The members have no conflict of interest. The approval will be applied for at the Scientific Ethics Committee Northern Region of Denmark. The study protocol will be registered in ClinicalTrial.gov and in the Region North Denmark.

   17. Compensation scheme information Not relevant for this project.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically verified prostate or rectal adenocarcinoma
2. Commenced to start curative EBRT to the pelvis, with or without chemotherapy or with or without androgen deprivation therapy (ADT)
3. Performance status 0-1
4. ≥ 18 years of age
5. Understanding and acceptance of written and orally informed consent in Danish

Exclusion Criteria:

1. Earlier treated with EBRT or other type of radiation to the pelvis
2. History of diagnosed inflammatory bowel disease
3. Colostomy
4. Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with curative EBRT for prostate or rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Frequency and classification of radiation-induced diarrhrea in patients with prostate and rectal cancer during curative external radiotherapy | 1 June 2022 - 31 December 2023
  Frequency of RID measured as mean number of stools per day/week, distribution daytime/night-time during EBRT.
  RID measured as Common Terminology Criteria (CTCAE)/Bristol Stool Scale (diarrhoea, rectal haemorrhage, bloating, abdominal pain, tenesmus, proctitis, rectal fissure, mucus, flatulence and faecal incontinence), score and use of antidiarrheal medication and laxatives (type, dose, start, stop).
  QoL measured during and following EBRT. Patient's nutrition, physical activity, biochemical measures and faecal samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, North Region, Denmark

REFERENCES:
- [Background] McBride WH, Schaue D. Radiation-induced tissue damage and response. J Pathol. 2020 Apr;250(5):647-655. doi: 10.1002/path.5389. Epub 2020 Feb 21. PMID 31990369
- [Background] Andreyev J. Gastrointestinal symptoms after pelvic radiotherapy: a new understanding to improve management of symptomatic patients. Lancet Oncol. 2007 Nov;8(11):1007-17. doi: 10.1016/S1470-2045(07)70341-8. PMID 17976611
- [Background] Muls AC. Acta Oncologica Lecture. Gastrointestinal consequences of cancer treatment and the wider context: a bad gut feeling. Acta Oncol. 2014 Mar;53(3):297-306. doi: 10.3109/0284186X.2013.873140. Epub 2014 Jan 27. PMID 24460087
- [Background] Morris KA, Haboubi NY. Pelvic radiation therapy: Between delight and disaster. World J Gastrointest Surg. 2015 Nov 27;7(11):279-88. doi: 10.4240/wjgs.v7.i11.279. PMID 26649150
- [Background] Stacey R, Green JT. Radiation-induced small bowel disease: latest developments and clinical guidance. Ther Adv Chronic Dis. 2014 Jan;5(1):15-29. doi: 10.1177/2040622313510730. PMID 24381725
- [Background] Andreyev HJ, Davidson SE, Gillespie C, Allum WH, Swarbrick E; British Society of Gastroenterology; Association of Colo-Proctology of Great Britain and Ireland; Association of Upper Gastrointestinal Surgeons; Faculty of Clinical Oncology Section of the Royal College of Radiologists. Practice guidance on the management of acute and chronic gastrointestinal problems arising as a result of treatment for cancer. Gut. 2012 Feb;61(2):179-92. doi: 10.1136/gutjnl-2011-300563. Epub 2011 Nov 4. PMID 22057051
- [Background] Khalid U, McGough C, Hackett C, Blake P, Harrington KJ, Khoo VS, Tait D, Norman AR, Andreyev HJ. A modified inflammatory bowel disease questionnaire and the Vaizey Incontinence questionnaire are more sensitive measures of acute gastrointestinal toxicity during pelvic radiotherapy than RTOG grading. Int J Radiat Oncol Biol Phys. 2006 Apr 1;64(5):1432-41. doi: 10.1016/j.ijrobp.2005.10.007. PMID 16580497
- [Background] Barnett GC, De Meerleer G, Gulliford SL, Sydes MR, Elliott RM, Dearnaley DP. The impact of clinical factors on the development of late radiation toxicity: results from the Medical Research Council RT01 trial (ISRCTN47772397). Clin Oncol (R Coll Radiol). 2011 Nov;23(9):613-24. doi: 10.1016/j.clon.2011.03.001. Epub 2011 Apr 5. PMID 21470834
- [Background] O'Brien PC, Franklin CI, Poulsen MG, Joseph DJ, Spry NS, Denham JW. Acute symptoms, not rectally administered sucralfate, predict for late radiation proctitis: longer term follow-up of a phase III trial--Trans-Tasman Radiation Oncology Group. Int J Radiat Oncol Biol Phys. 2002 Oct 1;54(2):442-9. doi: 10.1016/s0360-3016(02)02931-0. PMID 12243820
- [Background] Lawrie TA, Green JT, Beresford M, Wedlake L, Burden S, Davidson SE, Lal S, Henson CC, Andreyev HJN. Interventions to reduce acute and late adverse gastrointestinal effects of pelvic radiotherapy for primary pelvic cancers. Cochrane Database Syst Rev. 2018 Jan 23;1(1):CD012529. doi: 10.1002/14651858.CD012529.pub2. PMID 29360138
- [Background] Murphy J, Stacey D, Crook J, Thompson B, Panetta D. Testing control of radiation-induced diarrhea with a psyllium bulking agent: a pilot study. Can Oncol Nurs J. 2000 Summer;10(3):96-100. doi: 10.5737/1181912x10396100. PMID 11894282
- [Background] Itoh Y, Mizuno M, Ikeda M, Nakahara R, Kubota S, Ito J, Okada T, Kawamura M, Kikkawa F, Naganawa S. A Randomized, Double-Blind Pilot Trial of Hydrolyzed Rice Bran versus Placebo for Radioprotective Effect on Acute Gastroenteritis Secondary to Chemoradiotherapy in Patients with Cervical Cancer. Evid Based Complement Alternat Med. 2015;2015:974390. doi: 10.1155/2015/974390. Epub 2015 Nov 26. PMID 26693248
- [Background] Wedlake LJ, McGough C, Shaw C, Klopper T, Thomas K, Lalji A, Dearnaley DP, Blake P, Tait D, Khoo VS, Andreyev HJ. Clinical trial: Efficacy of a low or modified fat diet for the prevention of gastrointestinal toxicity in patients receiving radiotherapy treatment for pelvic malignancies. J Hum Nutr Diet. 2012 Jun;25(3):247-59. doi: 10.1111/j.1365-277X.2012.01248.x. Epub 2012 Apr 20. PMID 22515941
- [Background] Stryker JA, Bartholomew M. Failure of lactose-restricted diets to prevent radiation-induced diarrhea in patients undergoing whole pelvis irradiation. Int J Radiat Oncol Biol Phys. 1986 May;12(5):789-92. doi: 10.1016/0360-3016(86)90037-4. PMID 3086261
- [Background] Ravasco P, Monteiro-Grillo I, Vidal PM, Camilo ME. Dietary counseling improves patient outcomes: a prospective, randomized, controlled trial in colorectal cancer patients undergoing radiotherapy. J Clin Oncol. 2005 Mar 1;23(7):1431-8. doi: 10.1200/JCO.2005.02.054. Epub 2005 Jan 31. PMID 15684319
- [Background] Kozelsky TF, Meyers GE, Sloan JA, Shanahan TG, Dick SJ, Moore RL, Engeler GP, Frank AR, McKone TK, Urias RE, Pilepich MV, Novotny PJ, Martenson JA; North Central Cancer Treatment Group. Phase III double-blind study of glutamine versus placebo for the prevention of acute diarrhea in patients receiving pelvic radiation therapy. J Clin Oncol. 2003 May 1;21(9):1669-74. doi: 10.1200/JCO.2003.05.060. PMID 12721240
- [Background] Rotovnik Kozjek N, Kompan L, Soeters P, Oblak I, Mlakar Mastnak D, Mozina B, Zadnik V, Anderluh F, Velenik V. Oral glutamine supplementation during preoperative radiochemotherapy in patients with rectal cancer: a randomised double blinded, placebo controlled pilot study. Clin Nutr. 2011 Oct;30(5):567-70. doi: 10.1016/j.clnu.2011.06.003. Epub 2011 Jul 5. PMID 21733605
- [Background] Vidal-Casariego A, Calleja-Fernandez A, de Urbina-Gonzalez JJ, Cano-Rodriguez I, Cordido F, Ballesteros-Pomar MD. Efficacy of glutamine in the prevention of acute radiation enteritis: a randomized controlled trial. JPEN J Parenter Enteral Nutr. 2014 Feb;38(2):205-13. doi: 10.1177/0148607113478191. Epub 2013 Mar 7. PMID 23471208
- [Background] Kavanagh BD, Pan CC, Dawson LA, Das SK, Li XA, Ten Haken RK, Miften M. Radiation dose-volume effects in the stomach and small bowel. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S101-7. doi: 10.1016/j.ijrobp.2009.05.071. PMID 20171503
- [Background] Abbott J, Teleni L, McKavanagh D, Watson J, McCarthy AL, Isenring E. Patient-Generated Subjective Global Assessment Short Form (PG-SGA SF) is a valid screening tool in chemotherapy outpatients. Support Care Cancer. 2016 Sep;24(9):3883-7. doi: 10.1007/s00520-016-3196-0. Epub 2016 Apr 19. PMID 27095352
- [Background] Jager-Wittenaar H, Ottery FD. Assessing nutritional status in cancer: role of the Patient-Generated Subjective Global Assessment. Curr Opin Clin Nutr Metab Care. 2017 Sep;20(5):322-329. doi: 10.1097/MCO.0000000000000389. PMID 28562490
- [Background] Ottery FD. Definition of standardized nutritional assessment and interventional pathways in oncology. Nutrition. 1996 Jan;12(1 Suppl):S15-9. doi: 10.1016/0899-9007(96)90011-8. PMID 8850213